CLINICAL TRIAL: NCT06305351
Title: A 42-Day Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of K-757 And K-833 in Overweight/Obese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of K-757 and K-833 in Overweight/Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-757 P008
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- K-757 and K-833 combination (Experimental)
  Interventions: Drug: K-757 and K-833 QD; Drug: K-757 and K-833 BID
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757 and K-833 QD; Drug: Matching placebo to K-757 and K-833 BID

INTERVENTIONS:
Drug: K-757 and K-833 QD — Both administered orally once daily
  Arms: K-757 and K-833 combination
Drug: K-757 and K-833 BID — Both administered orally twice daily
  Arms: K-757 and K-833 combination
Drug: Matching placebo to K-757 and K-833 QD — Both administered orally once daily
  Arms: Placebo
Drug: Matching placebo to K-757 and K-833 BID — Both administered orally twice daily
  Arms: Placebo

SUMMARY:
This is a multiple dose study to evaluate the safety, tolerability, PK, and PD of K-757 and K-833 when co-administered in overweight/obese patients with Type 2 diabetes mellitus (T2DM)

ELIGIBILITY:
Inclusion Criteria:

1. Understand the trial procedures and agree to participate by providing written informed consent.
2. Be willing and able to comply with all trial procedures and restrictions, including following study diet requirements.
3. Be between 18 to 70 years of age, inclusive, at the Screening Visit.
4. Has T2DM in accordance with American Diabetes Association (ADA) guidelines at the Screening Visit.
5. Is on stable metformin monotherapy (total daily dose of 1,000 to 2,000 mg/day) for at least 3 months and tolerating metformin well in the opinion of the investigator. Note: Both the immediate release (IR) and extended release (XR) formulations of metformin are acceptable.
6. HbA1c of ≤7.5% at Screening.
7. Have a Body Mass Index (BMI) ≥25.0 and <40.0 (kg/m2) at the Screening Visit.
8. Be weight stable (<5% variation) over the last 3 months, by subject report.
9. Be a nonsmoker who has not used tobacco or nicotine-containing products (e.g. nicotine patch, e-cigarettes, vapes) for at least 3 months before administration of the initial dose of trial drug and agrees to abstain from smoking tobacco or the use of nicotine-containing products while on study.
10. Be judged to be in generally good health by the Investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead ECG, and vital sign measurements performed at the Screening Visit and before administration of the initial dose of trial drug.
11. Meet the following requirements:

    1. Is a male who agrees to all of the following:

       * If partner is a non-pregnant female of child-bearing potential: To use an appropriate method of contraception, including a condom with spermicidal cream or jelly, from the first dose of study drug until 14 days after the last dose of study drug. A male subject who has had a vasectomy procedure must use a condom but is not required to use spermicidal cream or jelly.
       * If partner is pregnant, to use a condom. Note: Contraception/condom requirements are waived if partner is NOT of child-bearing potential (i.e. is male or is a female who is post-menopausal or surgically sterile [post-hysterectomy, post-bilateral oophorectomy, and/or post-bilateral salpingectomy]).
       * To not donate sperm from the first dose of study drug until 14 days after the last dose of study drug.

       OR
    2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:

       * Postmenopausal (aged >45 years and with a minimum of 12 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level in the menopausal range as established for the laboratory performing the test.
       * Post hysterectomy, bilateral oophorectomy or bilateral salpingectomy, based on the subject's recall of their medical history.

       OR
    3. Is a female of reproductive potential and:

       * agrees to not donate eggs from the first dose of study drug until 14 days after the last dose of study drug
       * agrees to remain abstinent from heterosexual activitya or
       * agrees to use (or have their partner use) a birth control method that is highly effective and has low user dependency. Acceptable methods of birth control are:

         * Progestogen-only implant (e.g. etonogestrel implant)
         * Intrauterine device (IUD)
         * Intrauterine hormone-releasing system (IUS)
         * Bilateral tubal occlusion
         * Vasectomized partner a Abstinence can be used as the sole method of contraception if it is in line with the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ethics committees. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Has participated in another interventional investigational study within 30 days of the Screening Visit. The window will be derived from the date of the last study procedure and/or AE related to the study procedure in the previous study to the Screening Visit of the current study. If the subject received an investigational medication in the prior study, at least 5 half-lives (or longer if required by local regulations) must have passed between the last dose of the investigational product and the Screening Visit.
2. Is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the Sponsor or study site.
3. Has a history of multiple significant and/or any severe allergies (eg, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
4. Has a known hypersensitivity or contraindication to any component of K-757, K-833, including excipients.
5. Has a positive alcohol or drug screen at Screening or admission.
6. Has a positive pregnancy test.
7. Is a lactating/nursing female.
8. Has a positive test result for hepatitis B surface antigen (Ag), hepatitis C virus antibody, or human immunodeficiency (HIV) antibody, at the Screening Visit. Note: Subjects with positive hepatitis B virus or hepatitis C virus serology may be enrolled if quantitative polymerase chain reaction for hepatitis B virus or hepatitis C virus ribonucleic acid is negative.
9. Does not meet study site COVID-19 admission/study participation restrictions.
10. Has a fever (>38°C)*
11. Had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit*
12. Is unable to refrain from the use of prohibited prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication through completion of study participation.
13. Allowable concomitant medications may include 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins), ≤2 permissible anti-hypertensive agents, postmenopausal hormone replacement therapy (HRT), and/or proton pump inhibitors (PPIs).
14. Has been on any GLP-1 receptor agonist, any dipeptidyl peptidase IV (DPP-4) inhibitor, or any approved or investigational medications known to cause weight loss in the prior 3 months.
15. Has a history of type 1 diabetes mellitus (T1DM) or a history of diabetic ketoacidosis or subject assessed by the investigator as possibly having T1DM.
16. Has a history of other specific types of diabetes (e.g. genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post organ transplant diabetes).
17. Has been treated with insulin or any other anti-hyperglycemic agents (AHAs) other than metformin within 4 weeks of screening or within 12 weeks of screening if the AHA was a thiazolidinedione (e.g., rosiglitazone, pioglitazone).
18. At Screening or Day 1 has a site fasting fingerstick glucose of >270 mg/dL. If the Day -1 fasting fingerstick glucose is >270 mg/dL, a re-test may be conducted the morning of Day1 in fasted state prior to randomization. If the result is ≤270 mg/dL, the subject may be randomized if all other entry criteria are met.
19. Has evidence or history of diabetic complications or significant end organ damage, eg, proliferative retinopathy and/or macular edema, eGFR Modification of Diet in Renal Disease (MDRD) ≤60 mL/min, diabetic neuropathy.
20. One or more self-reported episodes of hypoglycemia (fingerstick glucose <60 mg/dL with symptoms consistent with hypoglycemia or <50 mg/dL irrespective of symptoms) within the last 3 months.
21. Is using or anticipates the need for using concomitant medications which are inhibitors of P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) or any prohibited medications listed in Section 10.1 from screening until the post study visit.
22. Has excessive consumption of alcohol within 6 months prior to screening (>14 drinks/week for men and >7 drinks/week for women, where l drink= 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) or any use of soft drugs (such as marijuana or any substances containing tetrahydrocannabinol (THC) or cannabidiol (CBD)) within 3 months prior to Screening, or hard drugs (such as cocaine) within 6 months prior to Screening.
23. Is unwilling or unable to refrain from consuming alcohol from 7 days prior to the first dose of study medication through the completion of study participation.
24. Has a substance abuse disorder.
25. Had a previous major psychotic disorder.
26. Has a corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec) for males and >470 msec for females at screening or admission.
27. Has a mean value for triplicate semi-recumbent systolic blood pressure >160 millimeters of mercury (mmHg) and/or diastolic blood pressure (BP) >95 mmHg measured after at least 10 minutes at rest at the Screening Visit. Note: If a subject's BP is exclusionary on the first triplicate assessment at the Screening visit, they may have 1 repeat triplicate BP assessment at that visit, after another rest of at least 10 minutes, to qualify for the study.

    If a subject's BP is exclusionary at screening but the investigator feels that BP is likely to be below the exclusionary thresholds at admission (Day -1), this criterion can be re-assessed at admission. Adjustment of doses of anti-hypertensives already being taken at screening is permissible, but initiation of new agents is not permissible. For subjects whose BP is exclusionary at Screening and at the first triplicate assessment on Day -1, triplicate assessments can be repeated up to twice on Day -1, as needed.

    Triplicate assessments should occur after a rest of at least 10 min. Also, the first measurement of any triplicate assessment should be separated from the last measurement in a prior triplicate assessment by at least 10 minutes.
28. Has alanine aminotransferase or aspartate aminotransferase (ALT or AST) of >1.5X upper limit of normal (ULN) or total bilirubin >1.5X ULN (isolated bilirubin >1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin is within the laboratory normal range) at Screening or admission. (Note: Subjects who do not meet this criterion at Screening or at admission may not be rescreened/retested).
29. Has serum amylase or lipase >1.2X the ULN at the Screening Visit.
30. Has a recent history (within past 3 years) or current diagnosis of any of the following GI (gastro-intestinal) related diseases: intestinal obstruction, GI perforation, GI motility disorders, adhesions, Clostridium difficile colitis or have had recent unexplained GI bleeding within 3 months prior to screening.
31. Has any history of pancreatitis (acute or chronic), gastroparesis, ischemic colitis, inflammatory bowel disease (IBD), celiac disease, irritable bowel syndrome (IBS), or colitis.
32. Has any past surgical history of gastric banding or bariatric surgery or bowel resection.
33. Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, neurologic disorder, neoplastic, or genitourinary abnormalities or diseases.
34. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

note* Subject may be included if they are able to return to the site within 7 days of initial screening and the exclusion criterion is no longer met.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who experienced 1 or more treatment-emergent AEs | Up to Day 43 +/- 2 days
Proportion of participants who discontinued study medication due to an AE | Up to Day 43 +/- 2 days

SECONDARY OUTCOMES:
Area under the concentration-time curve [AUC] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
AUC of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757
Maximum concentration [Cmax] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
Cmax of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757
Time of maximum concentration [Tmax] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
Tmax of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757
Clearance [Cl] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
Cl of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757
Volume of distribution at steady-state [Vdss] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
Vdss of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757
Half-life [t1/2] of plasma K-757 | Days 1, 28, 42
  when co-administered with K-833
t1/2 of plasma K-833 | Days 1, 28, 42
  when co-administered with K-757

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Miami, Miami, Florida, United States